CLINICAL TRIAL: NCT07262801
Title: Evaluating the Psychological and Physiological Impact of a Mindfulness-based Intervention on Anxiety Disorders During the Postpartum Period: A Proof of Concept Trial
Brief Title: Psychological and Physiological Impact of a Mindfulness-based Intervention on Anxiety Disorders During the Postpartum Period
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Sheryl Green, Dr. Sheryl Green, Ph.D., C.Psych, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPA-Mindfulness-RCT
Record Dates: First submitted 2025-09-19; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Postpartum Anxiety; Anxiety Disorders
Keywords: postpartum anxiety; anxiety disorders; mothers; mindfulness; mindfulness-based intervention; emotion regulation; interoception; fMRI; resting state functional connectivity
MeSH Terms: conditions — Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4-week mindfulness intervention (Experimental)
  Interventions: Behavioral: 4-week mindfulness-based intervention
- Waitlist treatment as usual control (No Intervention)

INTERVENTIONS:
Behavioral: 4-week mindfulness-based intervention — This is the first mindfulness-based intervention specifically designed for postpartum mothers and birthing parents with clinical anxiety. The protocol is adapted from Mindfulness-Based Cognitive Therapy for Depression (by J. Mark G. Williams, John D. Teasdale, and Zindel Segal), and is explicitly tailored to address anxiety disorders during the postpartum period. Most existing mindfulness-based protocols primarily target anxiety during pregnancy, are suitable for both clinical and subclinical levels of anxiety, and are commonly applied to both postpartum depression and anxiety populations.
  Arms: 4-week mindfulness intervention

SUMMARY:
Postpartum anxiety (PPA) affects up to 20% of mothers in the first year after delivery, with mothers often reporting both psychological and physical symptoms. Present non-pharmacological interventions are effective at improving some psychological aspects of PPA such as anxiety, depressive mood, and distress. However, current interventions are not effective in improving emotion regulation (ER), something that many with PPA experience impairment in. Current interventions also seldom target the physical aspects of anxiety, such as bodily awareness - sensing and understanding internal signals in the body (e.g., sensing a fast heartbeat). There is a link between ER and bodily awareness, however psychological interventions that target both these aspects have not been investigated in the PPA population. As a result, a mind-body intervention targeting both ER and bodily awareness is needed to offer a more holistic treatment option.

The purpose of the proposed study is to test the effectiveness of a 4-week mindfulness intervention on anxiety symptoms, ER, and bodily awareness in those with PPA. We will use self-report questionnaires alongside brain imaging (functional magnetic resonance imaging; fMRI) to evaluate the effectiveness. Combining both subjective and objective measures will provide greater confidence in our findings, ensuring a more comprehensive understanding of the intervention's impact. Self-report questionnaires will be administered at enrolment, immediately post-intervention, and 4 weeks post-intervention. Brain imaging will be conducted at enrolment and immediately post-intervention. We believe this intervention will lead to improvements in anxiety symptoms, ER, and bodily awareness on the questionnaires and fMRI scans.

If effective, the proposed mindfulness intervention will target a broader range of psychological and physical symptoms, and reduce the negative impact of PPA on mothers and their infants in Canada and beyond.

ELIGIBILITY:
Inclusion Criteria:

* mothers/birthing parents 18 years and older who are between 0-12 months postpartum
* principal diagnosis of an anxiety disorder as per the Diagnostic Assessment Research Tool (DART; Schneider et al., 2022), with or without comorbid depression
* no concurrent psychological treatment
* not taking psychoactive medication or a) medications are stable in dose and type for at least 8 weeks prior to the study (as per Canadian psychiatric guidelines; McQueen et al., 2016) and b) medications remain stable throughout the study
* fluent in English, minimal grade 8 reading level.

Exclusion Criteria:

* severe depression/suicidality requiring acute intervention
* women with psychotic or current alcohol or substance use disorders
* suffering from severe claustrophobia
* metallic objects in body (metal implants, pacemakers)
* currently pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
State-Trait Inventory for Cognitive and Somatic Anxiety (STICSA) | Administered at baseline (at enrolment), post-intervention (immediately after the 4 week intervention), and at the 3 months follow-up (3 months after intervention completion).

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) | Administered at baseline (at enrolment), post-intervention (immediately after the 4 week intervention), and at the 3 months follow-up (3 months after intervention completion).
Penn State Worry Questionnaire (PSWQ) | Administered at baseline (at enrolment), post-intervention (immediately after the 4 week intervention), and at the 3 months follow-up (3 months after intervention completion).
Generalized Anxiety Disorder 7-Item Scale (GAD-7) | Administered at baseline (at enrolment), post-intervention (immediately after the 4 week intervention), and at the 3 months follow-up (3 months after intervention completion).
Edinburgh Postnatal Depression Scale (EPDS) | Administered at baseline (at enrolment), post-intervention (immediately after the 4 week intervention), and at the 3 months follow-up (3 months after intervention completion).
World Health Organization Quality of Life Scale (WHOQoL) | Administered at baseline (at enrolment), post-intervention (immediately after the 4 week intervention), and at the 3 months follow-up (3 months after intervention completion).
Perceived Stress Scale (PSS) | Administered at baseline (at enrolment), post-intervention (immediately after the 4 week intervention), and at the 3 months follow-up (3 months after intervention completion).
Multidimensional Assessment of Interoceptive Awareness 2 (MAIA-2) | Administered at baseline (at enrolment), post-intervention (immediately after the 4 week intervention), and at the 3 months follow-up (3 months after intervention completion).
Interoceptive Sensitivity and Attention Questionnaire (ISAQ) | Administered at baseline (at enrolment), post-intervention (immediately after the 4 week intervention), and at the 3 months follow-up (3 months after intervention completion).
Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF) | Administered at baseline (at enrolment), post-intervention (immediately after the 4 week intervention), and at the 3 months follow-up (3 months after intervention completion).
Postpartum Bonding Questionnaire (PBQ) | Administered at baseline (at enrolment), post-intervention (immediately after the 4 week intervention), and at the 3 months follow-up (3 months after intervention completion).
Social Provisions Scale (SPS) | Administered at baseline (at enrolment), post-intervention (immediately after the 4 week intervention), and at the 3 months follow-up (3 months after intervention completion).
The Dyadic Adjustment Scale (DAS) | Administered at baseline (at enrolment), post-intervention (immediately after the 4 week intervention), and at the 3 months follow-up (3 months after intervention completion).

OTHER OUTCOMES:
Resting State Functional Connectivity (fMRI) | Completed at baseline (at enrolment) and post-intervention (immediately after the 4 week intervention), in participants randomized to the experimental group only.

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl M Green, Ph.D., C.Psych, Principal Investigator — St. Joseph's Healthcare Hamilton; Benicio N Frey, MD, PhD, FRCPC, Study Chair — St. Joseph's Healthcare Hamilton; Zoryana Babiy, M.Sc., Study Director — McMaster University
Locations (2):
- Canada (2):
  - Women's Health Concerns Clinic, St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Women's Health Concerns, St. Joseph's Healthcare Hamilton, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Experimental group participants will be given the option to consent to having their de-identified REDCap questionnaires and fMRI scans data shared with the Canadian Biomarker Integration Network in Depression (CAN-BIND). CAN-BIND is a standardized research platform that supports large-scale collaboration by collecting and curating data from both healthy and clinical populations. If one chooses to provide this optional consent, their data may be used to support future ethically approved research projects. All shared data will be encrypted and de-identified to protect privacy as CAN-BIND follows strict ethical and data security standards, comparable to those at St. Joseph's Healthcare Hamilton.
Supporting Information: ICF

REFERENCES:
- [Derived] Babiy Z, Frey BN, McCabe RE, Bieling PJ, Minuzzi L, Puccinelli C, Green SM. Mindfulness-Based Intervention for Treatment of Anxiety Disorders During the Postpartum Period: A 4-Week Proof-of-Concept Randomized Controlled Trial Protocol. Brain Sci. 2026 Jan 13;16(1):88. doi: 10.3390/brainsci16010088. PMID 41594809